CLINICAL TRIAL: NCT04895865
Title: A Comparison Between Two Repetition Prescription Approaches in Resistance Training Delivered Via Videoconferencing to Untrained Young Adults
Brief Title: Repetition Prescription Approaches Delivered Via Videoconferencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Israel Halperin, Senior faculty member, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHalperin
Record Dates: First submitted 2021-05-09; First posted 2021-05-20 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Health Behavior
Keywords: Physical activity; Exercise adherence; Resistance training; Affective responses; eHealth; Online exercise; Self-selection; Rating of Perceived Exertion
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention group receives alternative treatment Control group receives traditional treatment
Who Masked: Participant
Masking Description: Participants will be blinded to allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-selected (Experimental): Participants in the "self-selected" arm will choose the initial resistance in view of their preferences, and complete as many repetitions as they wish in order to reach the target rating of perceived exertion RPE of 7/10
  Interventions: Behavioral: RPE-based load and repetition number selection
- Predetermined (Active Comparator): Participants in the "predetermined" arm will be instructed to complete ten repetitions per set and exercise, while aiming to reach a rating of perceived exertion (RPE) of 7/10 by the 10th repetition. This means that participants will need to select and adjust the resistance of each exercise (e.g., band's resistance) to achieve this goal.
  Interventions: Behavioral: Predetermined load and number of repetitions

INTERVENTIONS:
Behavioral: RPE-based load and repetition number selection — Providing trainees with choices regarding the load and the number of repetitions to be performed per set and exercise
  Arms: Self-selected
Behavioral: Predetermined load and number of repetitions — Trainees predetermine the load and perform ten repetitions per set and exercise
  Arms: Predetermined

SUMMARY:
A randomized controlled trial comparing between two approaches of prescribing repetition-numbers in resistance training (RT) sessions on psychological, physiological, and performance outcomes. Sixty healthy and sedentary adults (age range: 18-45) will be randomly allocated to either the "predetermined" or "self-selected" groups. The groups will differ in the amount of choice they will be able to make concerning the resistance of each exercise and the number of repetitions they complete (see detailed description). Both groups will complete two sessions per week composed of body weight and resistance band exercises, lasting 45 minutes for eight weeks. The sessions will be delivered live by a certified instructor using a videoconferencing platform.

The primary aim of this study is:

Compare between the "predetermined" and the "self-selected" repetition prescription approaches on psychological, physiological, and performance outcomes in a cohort of 60 healthy and sedentary adults (age range: 18-45) over an eight-week period of live, videoconferencing RT sessions.

The secondary aim is:

Determine the influence of live, videoconferencing group RT sessions on psychological, physiological, and performance outcomes across groups.

DETAILED DESCRIPTION:
Background:

Providing trainees with more choices in exercise sessions is an autonomy supportive process which can lead to a more enjoyable experience, greater adherence to the training program and preferable performance outcomes. We will compare between two approaches to prescribing repetition-numbers in resistance training sessions- the "predetermined" and the "self-selected", based on the amount of choice trainees receive while training. Sixty healthy and sedentary adults (age range: 18-45) will train bi-weekly for 45 minutes using resistance bands in a live, videoconferencing group setting.

Intervention details:

The intervention will last eight weeks and include bi-weekly, 45-minute online sessions instructed by two alternating experienced instructors. Each session will include an introduction and setup (5-minutes), warm-up (5-minutes), body-weight and resistance band exercises (30-minutes) and cool down (5-minutes). We will upload the study protocol to an external server for more details.

Both groups will follow the exact same exercise program with one key difference: participants in the "predetermined" group will be instructed to complete 10 repetitions per set and exercise, while aiming to reach a rating of perceived exertion (RPE) of 7/10 by the 10th repetition. This means that participants will need to select and adjust the resistance of each exercise (e.g., band's resistance) to achieve this goal. Conversely, in the "self-selected" group, participants will choose the initial resistance in view of their preferences, and complete as many repetitions as they wish in order to reach the same target RPE of 7/10. Note that while the initial resistance, and thus, the number of repetitions is expected to differ between group, both are matched for perception of effort.

Recruitment and procedures:

Participants will be recruited via social media (i.e., Facebook Inc., Menlo Park, CA, USA). Each candidate will be screened for initial eligibility. After screening participants will be block-randomized to the "predetermined" of the "self-selected" groups, matched for age and gender. Participants will be blind to their allocation (see concealment section). Prior to visiting the exercise laboratory at Tel Aviv University for the testing session, participants will receive written materials regarding the exercise sessions, testing procedures, and the use of the Rating of Perceived Exertion (RPE) scale (0-10), and a video demonstrating the implementation of RPE in practice. All participants that are part of a given group will be required to complete the first testing session within a maximum of one week before the program begins, and the follow up testing session within a maximum of one week after the program ends. Practically, one group will begin and end all procedures (i.e., initial testing, eight-weeks program, follow up testing) one week before the other group. The order of which group will begin first will be randomly decided by a coin flip.

The initial testing session will include the following steps:

1. Sign an informed consent form.
2. Fill out the Basic Regulations in Exercise Questionnaire (BREQ).
3. Body composition analysis (see outcome measures section).
4. RPE terminology verification based on the videos and written materials delivered in advance.
5. Performance tests (see outcome measures section).
6. Practice how to use the resistance band (see below) and set up terminology to be used during the sessions (e.g. "open loop", "more tension").

That same order will be kept on the final tests (excluding the informed consent), which will also be conducted at the same place, at the same hour-window, and by the same experimenter.

Home-based equipment:

Participants will receive one elastic band (NT loops, purchased from: (https://www.ntloop.com/shop/) as they are affordable, accessible and allow exercising in a controlled, safe manner. When practicing with an elastic band, changing grip width, or rubber stiffness allows the trainee to achieve greater or lesser resistance.

Videoconferencing platform:

RT sessions will be delivered using "Zoom video communications" (San-Jose, CA, USA) due to its popularity and user-friendly interface. Additionally, a WhatsApp group chat (Facebook Inc., Menlo Park, CA, USA) will be created for each group to deliver updates and reminders. A technical assistant from the research team will be available during the live broadcast.

Sample size:

This sample size is based on our recruitment abilities and resources and based on our previous experience with this type of intervention. A sample size of 30 participants per group is considered large in exercise science research with both statistically and practically significant effects often detected. We also expect for future meta-analyses to take place and for this work to be included. Thus, even if this study is currently under-powered for small effects, it may add valuable data to the field of exercise science.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-active (characterized by 60 minutes or less per week of formal exercise sessions)
* Ages of 18-45
* Did not participate in RT in the past six months.
* Participants will be asked to fill out a health questionnaire. If they marked any of the items on the health questionnaire as positive (e.g., diabetes) they were asked to provide a medical clearance from a doctor.
* Signing a health declaration to participate in physical activity according to the government regulations

Exclusion Criteria:

* Orthopedic or neurological conditions
* Diagnosis of co-morbidities
* Routine use of prescription medication
* Pregnancy
* Less than six months after childbirth

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline enjoyment score | Change from week two to week four, week six and the end of the program on week eight.
  Participants will respond to a bi-monthly survey introducing the question: "how much did you enjoy the previous four sessions?" using a visual analog scale (VAS) ranging from (-100) (i.e., did not enjoy it at all) to 100 (i.e., enjoyed it very much). First, the change in scores from one time point the previous one will be calculated, resulting in three change scores across the duration of the study (e.g., week 4 minus week 2, week 6 minus week 4, etc.). Then, the three change scores will be averaged per group and compared between groups as the main outcome.

SECONDARY OUTCOMES:
Adherence proportion | Through study completion, a period of eight weeks.
  The proportion of adherence to the program calculated as session attended divided by the total sessions, times 100 over a period of eight weeks.
Change in fat free mass (FFM) | Change from baseline to the end of intervention at eight weeks.
  SECA mBCA 515 device (MFBIA; SECA®, Hamburg, Germany) will be used to measure bioimpedance. Participants will be asked to drink 400 ml of water on the day of measurement and up to 30 minutes before stepping on the feet-electrodes bare feet. Participants will hold the hand-electrodes and the flow of low alternating current will produce an output of FFM reported in units of kilograms.
Change in body mass index (BMI) | Change from baseline to the end of intervention at eight weeks.
  SECA mBCA 515 device (MFBIA; SECA®, Hamburg, Germany) will be used to measure body weight and height, which will be used to calculate BMI. Participants will be asked to stand on a stadiometer to measure their height, then step on the device which will measure their weight and produce an automated output of BMI score. The change in BMI from baseline to the end of the intervention will be used as a secondary outcome.
Change in maximal strength: | Change from baseline to the end of intervention at eight weeks.
  The isometric mid-thigh pull (IMTP) assesses maximal strength of the body's large muscle groups. Participants will pull a fixed bar while standing on force plates (Kinvent, Deltas force plates). The force plate will measure the mean force of the three-second test. Test units are kilograms.
Change in hand-grip strength: | Change from baseline to the end of intervention at eight weeks.
  The hand grip test assesses maximum strength of the grip muscles through squeeze the dynamometer (Kinvent, Grip dynamometer). Measurement units are kilogram, and the peak value will be used to calculate the change from baseline.
Change in knee-extensor strength: | Change from baseline to the end of intervention at eight weeks.
  The isometric knee extension test will measure force by a dynamometer device attached to a firm belt (Kinvent, Link pull dynamometer). Measurement units are kilogram, and the mean force will be used for analysis.
Change in lower-body explosive power: | Change from baseline to the end of intervention at eight weeks.
  The counter movement jump test assesses lower body explosive power using a force plate (Kinvent, Deltas force plates). Participants will stand on the force plate with their hands on their waist and jump as high as possible. The measurement unit is centimeter, and the peak value will be used for analysis.
Change in upper body endurance: | Change from baseline to the end of intervention at eight weeks.
  The push-up test assesses muscular endurance of the upper body muscle groups. Participants will perform the maximal number of push-ups with their body straight and their chest touching a target. Participants will use an inclination if they cannot complete five repetitions before beginning the test. Inclination height will be recorded. The number of repetitions will be used for analysis.
Change in perception of autonomy: | Change from week two to week four, week six and the end of the program on week eight.
  Participants will be presented with three questions concerning their perceived autonomy. Participants will be asked to rate their response on a Visual Analog Scale (VAS) ranging from (-100) (i.e., not autonomous at all) to 100 (extremely autonomous). First, the change in scores from one time point the previous one will be calculated, resulting in three change scores across the duration of the study (e.g., week 4 minus week 2, week 6 minus week 4, etc.). Then, the three change scores will be averaged per group and compared between groups as a secondary outcome.
Change in satisfaction with the program: | Change from week two to week four, week six and the end of the program on week eight.
  Participants will be presented with three questions concerning their satisfaction with the variety of exercises, the instructor and the resistance band. Participants will be asked to rate their response on a Visual Analog Scale (VAS) ranging from (-100) (i.e., not satisfied at all) to 100 (i.e, extremely satisfied). First, the change in scores from one time point the previous one will be calculated, resulting in three change scores across the duration of the study (e.g., week 4 minus week 2, week 6 minus week 4, etc.). Then, the three change scores will be averaged per group and compared between groups as a secondary outcome.
Change in response to the ease of use of the rating of perceived exertion (RPE) scale: | Change from week two to week four, week six and the end of the program on week eight.
  Participants will be presented with two questions concerning the use of the RPE scale during the sessions. Participants will be asked to rate their response on a Visual Analog Scale (VAS) ranging from (-100) (not easy to use) to 100 (very easy to use). The average score of the three items will be used for analysis.
Change in the satisfaction with technology: | Change from week two to week four, week six and the end of the program on week eight.
  Participants will be presented with two questions concerning the use of technology (videoconferencing interface) during the sessions. Participants will be asked to rate their response on a Visual Analog Scale (VAS) ranging from (-100) (i.e., not satisfied at all) to 100 (i.e., extremely satisfied). First, the change in scores from one time point the previous one will be calculated, resulting in three change scores across the duration of the study (e.g., week 4 minus week 2, week 6 minus week 4, etc.). Then, the three change scores will be averaged per group and compared between groups as a secondary outcome.
Change in Basic Regulation to Exercise Questionnaire (BREQ-3) score: | Change from baseline to the end of the intervention (up to seven days from the end of week eight).
  Participants will respond to a 24-items questionnaire. Items are designed to explore the underlying motives to engaging in physical activity. The Likert-based items range from 0 (i.e., not true for me) to 4 (i.e., very true for me). The total score of the questionnaire will be calculated for the baseline response at the beginning of the intervention and the final response at the end of the intervention, and compared between the two groups. The absolute change in scores will be used as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Halperin, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

REFERENCES:
- [Background] Schwartz H, Har-Nir I, Wenhoda T, Halperin I. Staying physically active during the COVID-19 quarantine: exploring the feasibility of live, online, group training sessions among older adults. Transl Behav Med. 2021 Mar 16;11(2):314-322. doi: 10.1093/tbm/ibaa141. PMID 33447852
- [Background] Patall EA, Cooper H, Robinson JC. The effects of choice on intrinsic motivation and related outcomes: a meta-analysis of research findings. Psychol Bull. 2008 Mar;134(2):270-300. doi: 10.1037/0033-2909.134.2.270. PMID 18298272
- [Background] Lopes JSS, Machado AF, Micheletti JK, de Almeida AC, Cavina AP, Pastre CM. Effects of training with elastic resistance versus conventional resistance on muscular strength: A systematic review and meta-analysis. SAGE Open Med. 2019 Feb 19;7:2050312119831116. doi: 10.1177/2050312119831116. eCollection 2019. PMID 30815258
- [Background] Emanuel A, Har-Nir I, Rozen Smukas II, Halperin I. The effect of self-selecting the number of repetitions on motor performance and psychological outcomes. Psychol Res. 2021 Sep;85(6):2398-2407. doi: 10.1007/s00426-020-01402-4. Epub 2020 Aug 10. PMID 32778961
- See also: Resistance bands used in the intervention — https://www.ntloop.com/shop/